CLINICAL TRIAL: NCT05226962
Title: The Effects of Acute Ketone Monoester Supplementation on 20-Minute Time-Trial Performance in Trained Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Martin Gibala, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13837
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Exercise; Ketosis
Keywords: Performance
MeSH Terms: conditions — Motor Activity; Ketosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone (Active Comparator): An acute bout of exercise performed after the ingestion of a commercial ketone monoester supplement.
  Interventions: Dietary Supplement: Ketone monoester
- Control (Placebo Comparator): An acute bout of exercise performed after the ingestion of a taste-matched placebo supplement.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone monoester — A commercial liquid supplement ingested in a dose intended to provide ~0.35 g of ketone monoester per kg body mass of the participant
  Arms: Ketone
Other: Placebo — A liquid placebo that is volume- and taste-matched to the ketone monoester supplement
  Arms: Control

SUMMARY:
Diet can alter blood ketone levels and this in turn may affect exercise capacity. This study will determine if the acute ingestion of a ketone supplement alters cycling time trial performance. Participants will perform two trials in a randomized order. Each trial will involve a 20-minute bout of cycling on a stationary ergometer. Participants will ingest either a ketone supplement or a taste-matched placebo drink prior to exercise. Blood samples will be obtained to assess selected metabolic responses. This study will provide information regarding the effect of ketone supplementation on exercise responses.

DETAILED DESCRIPTION:
This study will determine if the acute ingestion of a ketone supplement alters cycling time trial performance. Trained participants with competitive cycling experience will be recruited. Exercise will involve a 20-minute bout of cycling on a stationary ergometer with the goal of producing the highest power output possible. Participants will ingest either a ketone supplement or a taste-matched placebo drink prior to exercise using a randomized, double-blind crossover design. Diet prior to exercise will be standardized between trials for a given participant. Blood samples will be obtained to assess selected metabolic responses. This study will provide information regarding the effect of ketone supplementation on exercise responses.

ELIGIBILITY:
Inclusion Criteria:

* Habitually ingesting >50 g of dietary carbohydrate daily i.e. not following a ketogenic diet.
* Regularly performing cycling exercise at least 3 days per week and for a total of ≥5 hours per week.
* Having an estimated peak oxygen uptake of ≥55 ml/kg/min for males and ≥48 ml/kg/min for females based on the online fitness calculator available at: www.worldfitnesslevel.org.
* Having competitive cycling experience.

Exclusion Criteria:

- Experiencing a condition that might preclude safe participation in physical activity and exercise, as determined by answering "Yes" to any question on Page 1 of the Canadian Society for Exercise Physiology Get Active Questionnaire.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Power output | 20-minute measurement during exercise
  Mean power output produced while cycling

SECONDARY OUTCOMES:
Heart rate | 20-minute measurement during exercise
  Mean heart rate while cycling
Perceived exertion | Single measurement immediately after exercise
  Rating of perceived exertion while cycling
Blood ketone | Single measurement immediately prior to exercise
  Blood ketone before exercise
Blood glucose | 20-minute measurement during exercise
  Mean blood glucose while cycling

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gibala, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No